CLINICAL TRIAL: NCT00706862
Title: FORTIS-C: A Phase 3, Randomized, Placebo-controlled Study of Oral Talactoferrin in Combination With Carboplatin and Paclitaxel as First-line Therapy in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Safety and Efficacy of Talactoferrin in Addition to Standard Chemotherapy in Patients With Non-small Cell Lung Cancer
Acronym: FORTIS-C
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LF-0208
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; Talactoferrin; Dendritic cell recruiter and activator; DCRA; Immunomodulatory agent; Lactoferrin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — talactoferrin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Talactoferrin, Carboplatin, Paclitaxel
  Interventions: Drug: Talactoferrin
- 2 (Placebo Comparator): Placebo, Carboplatin, Paclitaxel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talactoferrin — Oral, 1.5 grams twice per day
  Other Names: talactoferrin alfa; TLF; recombinant human talactoferrin; rhLF
  Arms: 1
Drug: Placebo — Oral, twice per day
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether the combination of talactoferrin, carboplatin and paclitaxel improves progression free survival and overall survival in patients with non-small cell lung cancer compared to the combination of paclitaxel and carboplatin alone

ELIGIBILITY:
Inclusion Criteria:

* Confirmed locally advanced or metastatic non-small cell lung cancer that is unresectable
* At least 1 unirradiated target lesion measurable by RECIST
* Adequate hematologic, renal and hepatic function
* ECOG 0,1
* Able to understand and sign an Informed Consent

Exclusion Criteria:

* Presence of brain metastases, unless the patient received brain irradiation, including adequate stereotactic radiosurgery, at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 3 weeks prior to randomization
* Received prior systemic anti-cancer therapy for NSCLC
* History of allergic reactions to compounds of similar chemical or biologic composition to talactoferrin or the chemotherapy drugs
* Any gastrointestinal tract disease or other medical condition resulting in the inability to take oral medications
* History of other malignancies except: (i) adequately treated basal or squamous cell carcinoma of the skin; (ii) curatively treated, a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (iii) other curatively treated solid tumor with no evidence of disease for ≥5 years
* Uncontrolled ischemic heart disease, or uncontrolled symptomatic congestive heart failure
* Serious active infection
* Psychiatric illness/social situations that would limit study compliance
* Other uncontrolled serious chronic disease or conditions that in the investigator's opinion could render compliance or follow-up in the protocol problematic
* Concurrent radiotherapy or radiotherapy within 4 weeks prior to randomization or previous radiotherapy at the indicator sites (the sites that are to be followed for determination of a response)
* Concurrent systemic corticosteroid therapy within 4 weeks prior to randomization, except prophylactic use of steroids prior to paclitaxel administration
* Known HIV positive or on active anti-retroviral therapy
* Known Hepatitis B surface antigen positive or hepatitis C positive
* Receipt of any investigational medication within 4 weeks prior to randomization
* Pregnant or lactating patients, or fertile female patients with a positive pregnancy test, or fertile female patients unwilling to use adequate contraception during treatment and for 30 days after completion of treatment
* Sexually active male patients unwilling to practice contraception while participating on the study and up to 30 days after completion of treatment
* Legal incapacity or limited legal capacity, unless authorization is granted by a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2009-02; Primary Completion 2015-06 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | After the occurence of the required number of events
Progression free survival | At the time of final analysis

SECONDARY OUTCOMES:
Objective response and disease stabilization rate | At the time of final analysis
Safety and tolerability | At the time of final analysis

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - Rush University Medical Center, Chicago, Illinois
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee